CLINICAL TRIAL: NCT05258448
Title: The Effect of Radiotherapy on the Heart in Loco-regional Advanced NSCLC Patients Treated With Definitive Radiotherapy Measured by Cardiac MR
Brief Title: COr Loco-regional Advanced Lung Cancer Treated With Chemo-radiotherapy (COLA)
Acronym: COLA
Status: Recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Agon Olloni, Principal Investigator, MD, Phd Student, Odense University Hospital
Other Study IDs: S-20160086
Record Dates: First submitted 2022-02-03; First posted 2022-02-28 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Cardiac Toxicity; Lung Cancer Stage III; Lung Cancer Stage II; Radiation Toxicity; Cardiac Disease
MeSH Terms: conditions — Cardiotoxicity; Lung Neoplasms; Radiation Injuries; Heart Diseases | interventions — Chemoradiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COLA 1: Locally advanced non-small-cell lung cancer: Patients with locally advanced non-small-cell lung cancer treated with radiotherapy alone or in combination with chemotherapy with curative intent. Patients are included before initiation of the treatment. A Cardiac MR and ECG are performed at the beginning of the treatment, and at 6, 12, and 24 months after radiotherapy.
  Interventions: Other: Chemoradiotherapy
- COLA 2 Locally advanced non-small-cell lung cancer: Patients with locally advanced non-small-cell lung cancer treated with radiotherapy alone or in combination with chemotherapy with curative intent. Patients not included in COLA 1 cohort are offered one cardiac MR and ECG between 12-24 months after radiotherapy treatment.
  Interventions: Other: Chemoradiotherapy

INTERVENTIONS:
Other: Chemoradiotherapy — Cardiac Magnetic Resonance scan and ECG

SUMMARY:
Patients with loco-regional NSCLC planned for curative treatment with chemoradiotherapy will be invited to participate in a prospective study; besides routine treatment, the patients will be followed with an ECG and cardiac MR for at least two years after radiotherapy treatment.

DETAILED DESCRIPTION:
Definitive chemo-radiotherapy is the treatment of choice for loco-regional advanced non-small cell lung cancer (LA-NSCLC). However, the treatment is associated with a range of side effects with radiation pneumonitis and esophagitis. In addition, the toxicity of the heart in lung cancer patients treated with radiotherapy has been offered less consideration. Therefore, it is essential to investigate the possible early and late toxicity to the heart and the baseline cardiac status of these patients. This study will describe cardiac comorbidity before radiotherapy treatment by a thorough history. Furthermore, we will evaluate heart function and evaluate possible heart disease by an ECG and cardiac MR. Patients will be followed with ECG and cardiac MR for two years after radiotherapy, detecting structural changes caused by radiotherapy and subclinical disease after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 Years
* Inoperable and histologically/cytologically verified NSCLC.
* Planned treatment with curative intent.
* Capable of completing study procedures ECG and Cardiac MR.
* Able of giving written and informed consent before study procedures are initiated.

Exclusion Criteria:

* Vulnerable patients.
* Patients with operable devices as pacemaker/ICD and cochlear implant or other conditions where MR scan is contraindicated.
* Claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced non-small-cell lung cancer will be included at the department of oncology at Odense University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 Years
  All cause mortality
Change in Left Ventricular Ejection Fraction | Baseline, at 6, 12 and 24 months.
  Change from baseline, evaluated by cardiac MR
Number of participants with treatment related adverse events and cardiac disease after radiotherapy as assesed by CTCAE v4.0. | 2 years.
  Assesed by patient interview and review of medical record.
Cardiovascular specific mortality | 2 years.
  Assesed by patient interview and review of medical record

SECONDARY OUTCOMES:
Late enhacment | At Baseline, 6, 12 and 24 months.
  Evaluated by cardiac MR.
LVEDV changes | 2 years
  Left ventricular enddiastolic change in cMR
LVESV changes | 2 years
  Left ventricular endsystolic change in cMR
LV mass in gram | 2 years
  Left ventricular mass in gram.

CONTACTS AND LOCATIONS:
Overall Officials: Tine Schytte, Professor, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: Undecided